CLINICAL TRIAL: NCT04632316
Title: A Prospective Phase I/IIa, Open-label, Multicenter Trial to Evaluate the Safety and Efficacy of oNKord®, an Off-the-shelf, ex Vivo-cultured Allogeneic NK Cell Preparation, in Subjects With Acute Myeloid Leukemia Who Are in Morphologic Complete Remission With Measurable Residual Disease and Who Are Currently Not Proceeding to Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: A Trial to Evaluate the Safety and Efficacy of oNKord® in Subjects With Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glycostem Therapeutics BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WiNK; 2019-003686-17 (EudraCT Number)
Record Dates: First submitted 2020-11-02; First posted 2020-11-17 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; NK cells; Umbilical cord blood; oNKord; ATMP; Off the shelf; Cell therapy; Immunotherapy; Oncology; Leukemia; Blood cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms; Leukemia; Hematologic Neoplasms | interventions — CF regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oNKord® (Experimental): Allogeneic ex vivo-generated Natural Killer (NK) cells from CD34+ umbilical cord blood progenitor cells
  Interventions: Drug: Cyclophosphamide-Fludarabine (Cy/Flu); Drug: oNKord®

INTERVENTIONS:
Drug: Cyclophosphamide-Fludarabine (Cy/Flu) — Lymphodepleting conditioning regimen
Drug: oNKord® — Allogeneic ex vivo-generated Natural Killer (NK) cells from CD34+ umbilical cord blood progenitor cells

SUMMARY:
WiNK is a Phase I/IIa trial to evaluate the safety and efficacy of oNKord® in 33 adults with acute myeloid leukemia (AML) who are in morphologic complete remission with residual measurable disease and who are currently not proceeding to allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
WiNK is a prospective 2-stage, open-label, single arm, multicenter Phase I/IIa trial to evaluate the safety and efficacy of oNKord®, an off-the-shelf, ex vivo-cultured allogeneic NK cell preparation, in 33 adults with acute myeloid leukemia (AML) who are in morphologic complete remission (CR) with residual measurable disease (MRD) and who are currently not proceeding to allogeneic hematopoietic stem cell transplantation (allo-HSCT).

Following informed consent and eligibility procedures, subjects enrolled in the trial will receive a lymphodepleting conditioning regimen consisting of cyclophosphamide and fludarabine (Cy/Flu) followed by up to 3 oNKord® infusions 4 days apart.

Stage A of the trial (dose escalation stage) is designed to assess the safety and tolerability of up to 3 oNKord® infusions, 4 days apart, in 3 cohorts of 3 subjects, and to determine the oNKord® recommended Phase II dose (RP2D) to be used in Stage B.

Stage B of the trial (expansion stage) will evaluate the safety, tolerability and efficacy of oNKord® at the RP2D in 24 subjects.

All subjects treated with oNKord® will be followed up until 12 months after the start of treatment. Eligibility criteria for participation in the trial and follow-up duration are the same for subjects in both Stage A and Stage B.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years old
2. Subjects with a diagnosis of AML and related precursor neoplasms according to the WHO 2016 classification (excluding acute promyelocytic leukemia), including secondary AML after an antecedent hematological disease (e.g. myelodysplastic syndrome) and therapy-related AML
3. Subjects who have achieved morphologic CR, including CRi and complete clinical remission, with MRD documented at screening, as assessed by centralized MFC, after one or two courses of remission induction chemotherapy and who have completed consolidation chemotherapy or who achieved morphologic CR with documented MRD with hypomethylating agents or other relevant appropriate therapies
4. Subjects who are currently (at the time of screening) not proceeding to allo-HSCT
5. Life expectancy ≥ 6 months at screening
6. Adequate renal and hepatic functions within 14 days of study screening, unless clearly disease related, as indicated by the following laboratory values:

   1. Serum creatinine ≤ 3 times the upper limit of normal (ULN) and estimated glomerular filtration rate (eGFR) ≥ 30 ml/min/1.73m2
   2. Serum total bilirubin < 2.0 mg/dl, unless due to Gilbert's syndrome
   3. Alanine transaminase (ALT) ≤ 2.5 x ULN
7. Karnofsky Status ≥ 50%
8. Seropositivity for EBV
9. Male subjects with partners who are women of childbearing potential must use an effective contraceptive method during the trial and for a minimum of 6 months after trial treatment, or have undergone successful vasectomy at least 6 months prior to entry into the trial (confirmed by semen analysis).
10. Female subjects of childbearing potential must have a negative serum pregnancy test at screening and agree to use an effective contraceptive method during the trial and for a minimum of 6 months after trial treatment.
11. Able to understand and willing to provide written informed consent to participate in the trial
12. Affiliation to a national health insurance scheme (according to applicable local requirements)

Exclusion Criteria:

1. Subjects having received prior allogeneic HSCT
2. Subjects with acute promyelocytic leukemia
3. Diagnosis of any previous or concomitant malignancy is an exclusion criterion, except when the subject completed treatment (chemotherapy and/or surgery and/or radiotherapy) with curative intent for this malignancy at least 6 months prior to enrolment
4. Blast crisis of chronic myeloid leukemia
5. Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, uncontrolled hypertension, active or uncontrolled infection) including abnormal laboratory values, that could compromise compliance with the trial protocol or cause unacceptable safety risks
6. Known allergy to any of the components of oNKord® (e.g., dimethyl sulfoxide [DMSO]) or to any of the drugs to be administered in the preparative regimen to oNKord® infusion
7. Contraindication to any of the drugs to be administered in the conditioning regimen or oNKord® infusion. This includes Cy, Flu, and medications associated with prophylaxis of AEs
8. Cardiac dysfunction as defined by:

   1. Myocardial infarction within the last 3 months of trial entry, or
   2. Reduced left ventricular function with an ejection fraction < 40% as measured by multi-gated acquisition (MUGA) scan or echocardiogram (echo) within 28 days before screening, or
   3. Unstable angina, or
   4. New York Heart Association (NYHA) Class IV congestive heart failure, or
   5. Unstable cardiac arrhythmias
9. Pulmonary dysfunction as defined by oxygen saturation < 90% on room air. Pulmonary function test (PFT) is required only in the case of symptomatic or prior known impairments within 28 days before screening - with pulmonary function < 50% corrected diffusing capacity of the lung for carbon monoxide (DLCO) and forced expiratory volume in 1 second (FEV1)
10. Major surgery within 4 weeks prior to screening or a major wound that has not fully healed
11. Vaccination with live, attenuated vaccines within 4 weeks prior to screening
12. Immunosuppressive drugs for concomitant disease. Subject must be able to be off prednisone or other immunosuppressive medications for at least 3 days prior to the start of Cy/Flu regimen
13. History of stroke or intracranial hemorrhage within 6 months prior to screening
14. Active infections (viral, bacterial or fungal) that requires specific therapy. Acute anti-infectious therapy must have been completed within 14 days prior to trial treatment
15. History of human immunodeficiency virus (HIV) or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
16. Subjects who are undergoing or will be undergoing chemotherapy (including HMAs), radiation therapy, targeted therapy or immunotherapy that cannot be finished or stopped at least 1 week prior to initiating the Cy/Flu conditioning regimen
17. Positive pregnancy test or breastfeeding for women of childbearing potential
18. Use of other investigational drugs/therapies within 3 weeks prior to trial treatment (within 6 weeks in the case of drugs/therapies with long half-life) or participation in a concomitant interventional clinical trial
19. Any serious concomitant medical condition, medication or therapy which could, in the opinion of the Investigator, compromise participation in the trial
20. Subjects under legal protection measure (guardianship, trusteeship or safeguard of justice) and/or inability or unwillingness to comply with the requirements and procedures of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of oNKord® using the cumulative incidence of the adverse events of special interest (AESI) | Up to 12 months
  AESI include: Grade 3 to 4 infusion-related toxicity of oNKord®, as rated by CTCAE v5.0; Acute GVHD grade III and IV; CRS and ICANS ≥ Grade 2, as rated by the ASTCT Consensus Grading
Efficacy of oNKord® using the cumulative incidence of MRD response as assessed by centralized assessment in bone marrow | Up to 12 months
  Subjects with responses are defined as MRD negative subjects still in morphologic CR at any time during the follow-up period of the trial after receiving oNKord® at RP2D

SECONDARY OUTCOMES:
Safety and tolerability of the overall trial treatment (Cy/Flu in combination with up to three oNKord® infusions) using the cumulative incidence of AESI | Up to 12 months
  AESI include: Grade 3 to 4 infusion-related toxicity of oNKord® as rated by CTCAE v5.0; Acute GVHD grade III and IV; CRS and ICANS ≥ Grade 2 as rated by the ASTCT Consensus Grading; Hemorrhagic cystitis; Death related to the overall trial treatment; Incidence and severity of viral, fungal, and bacterial infections with onset during the first two months following conditioning initiation, including viral reactivations, and infection related mortality defined as death due to infectious disease
Efficacy of the overall trial treatment (Cy/Flu in combination with oNKord® at RP2D) on event-free survival (EFS) | Up to 12 months
Efficacy of the overall trial treatment (Cy/Flu in combination with oNKord® at RP2D) on cumulative incidence of relapse (CIR) | Up to 12 months
Efficacy of the overall trial treatment (Cy/Flu in combination with oNKord® at RP2D) on the duration of MRD response | Up to 12 months
Efficacy of the overall trial treatment (Cy/Flu in combination with oNKord® at RP2D) on overall survival (OS) | Up to 12 months
Changes in Quality of Life (EORT QLQ-C30) | Up to 12 months
Changes in Quality of Life (SF-36) | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Arnold Ganser, MD, Principal Investigator — Hannover Medical School (MHH), Hannover, Germany
Locations (10):
- Belgium (2):
  - University Hospital Ghent, Ghent
  - University Hospital Leuven, Leuven
- Institut Gustave Roussy, Villejuif, France
- Germany (4):
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Hannover Medical School, Hanover
  - University Hospital Mainz, Mainz
- Amsterdam UMC, Amsterdam, Netherlands
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raimo M, Zavoianu AG, Meijs W, Scholten P, Spanholtz J. Qualification of a flow cytometry-based method for the evaluation of in vitro cytotoxicity of GTA002 natural killer cell therapy. Heliyon. 2024 Jan 17;10(2):e24715. doi: 10.1016/j.heliyon.2024.e24715. eCollection 2024 Jan 30. PMID 38304826